CLINICAL TRIAL: NCT02144155
Title: Open-label Study of the Long-Term Efficacy of Intranasal Oxytocin in Patients With Schizophrenia
Brief Title: Open-label Study of the Efficacy of Intranasal Oxytocin in Schizophrenia
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Break in funding
Sponsor: University of California, San Diego (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 120005
Record Dates: First submitted 2014-05-19; First posted 2014-05-21 (Estimated); Results first posted 2019-12-09 (Actual); Last update posted 2019-12-09 (Actual); Status verified 2019-12

CONDITIONS: Schizophrenia
Keywords: Oxytocin
MeSH Terms: conditions — Schizophrenia | interventions — Oxytocin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Oxytocin: 24 IU - 168 IU (Experimental): Oxytocin twice daily for 3 weeks
  Interventions: Drug: Oxytocin: 24IU - 168 IU
- Vehicle placebo (Sham Comparator): Placebo for 3 weeks
  Interventions: Drug: Oxytocin: 24IU - 168 IU; Drug: Placebo

INTERVENTIONS:
Drug: Oxytocin: 24IU - 168 IU — Oxytocin: 24IU - 168 IU
Drug: Placebo — placebo drug
  Arms: Vehicle placebo

SUMMARY:
The Objective of this study is to investigate the long-term efficacy of intranasal oxytocin in improvement of symptoms in patients with schizophrenia who have residual symptoms dispute being on adequate treatment with antipsychotic medication.

DETAILED DESCRIPTION:
Approximately 20 patients will be enrolled to participate in a 6 month flexible dose of oxytocin.

ELIGIBILITY:
Inclusion Criteria:

1. Adult men or women, 18 years of age or older.
2. Meet DSM-IV criteria for Schizophrenia
3. Women of childbearing potential must test negative for pregnancy at the time of enrollment based on urine pregnancy test and agree to use a reliable method of birth control during the study.
4. Must be on a therapeutic dose of 1 or 2 atypical antipsychotic medications (examples but not limited to Clozapine Olanzapine, Risperidone, Ziprasidone, Aripiprazole, Seroquel) with no major dose changes for at least 4 weeks.
5. A minimum PANSS total score of 55 at baseline and a score of at least 4 (moderate) on the subscale of the PANSS (suspiciousness/persecution) at screening.
6. Have a Clinical Global Impressions-Severity (CGI-S) scale score of at least 4 (moderately ill) at baseline;
7. Must be able to communicate effectively with the investigator and study coordinator and have the ability to provide informed consent.
8. Must be able to use nasal spray
9. Must demonstrate an acceptable degree of compliance with medication and procedures in the opinion of the investigator.

Exclusion Criteria:

1. Are pregnant or are breastfeeding (negative pregnancy test at screening)
2. A urine drug screen performed at screening must not show evidence of recent use of drugs of abuse
3. Any active medical condition that in the opinion of the investigator will interfere with the objectives of the study
4. Are unsuitable in any way to participate in this study, in the opinion of the investigator.
5. Another current, primary DSM-IV diagnosis other than Schizophrenia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2012-03 (Actual); Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- UCSD Medical Center - Hillcrest, San Diego, California, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- All Participants: This study was halted due to an indefinite break in funding. The Principal Investigator has left the institution and there is no way to determine the arms/groups of this study.
Period: Overall Study
Arm/Group | All Participants
Started | 14
Completed | 14
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | All Participants
Number analyzed (Participants) | 14
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: The PI has left the institution and this study was terminated due to loss of funding. The age of the participants enrolled cannot be located.
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 7
  White | 5
  More than one race | 0
  Unknown or Not Reported | 2

OUTCOME MEASURES:

1. Primary Outcome: Change in Total Score in the Positive and Negative Syndrome Scale (PANSS) From Baseline to 28 Weeks
Description: The three subscales of the PANSS include the Positive scale (7 items), the Negative scale (7 items), and the General Psychopathology scale (16 items). The total PANSS score is the sum of all 30 items of which each item is scored on a 1-7 rating system (7 indicating the worst symptoms). The items on the PANSS focus on symptoms that are common in patients with psychotic disorders and include hallucinations, delusions and disorganization as well as mood disturbances.
Time Frame: baseline and 28 weeks
Population: The PI has left the institution and this study was terminated due to loss of funding. The data was not analyzed.
Arm/Group | All Participants
Number analyzed (Participants) | 0

2. Secondary Outcome: Global Assessment of Functioning (GAF)
Description: The GAF considers psychological, social, and occupational functioning on a hypothetical continuum of mental health illness. Scores on the GAF range from 1 (extremely severe) to 100 (superior functioning).
Time Frame: 28 weeks
Population: The PI has left the institution and this study was terminated due to loss of funding. The data was not analyzed.
Arm/Group | All Participants
Number analyzed (Participants) | 0

3. Secondary Outcome: Clinical Global Impression-Severity
Description: The CGI-S is used to evaluate changes in overall severity of illness. Scores range from 1 (not at all) to 7 (among the most extremely ill).
Time Frame: 28 Weeks
Population: The PI has left the institution and this study was terminated due to loss of funding. The data was not analyzed.
Arm/Group | All Participants
Number analyzed (Participants) | 0

4. Secondary Outcome: Clinical Global Impression-Global Improvement (CGI-I)
Description: The CGI-I is a global assessment to evaluate the subject's improvement or worsening from baseline. Scores on the CGI-I scale range from 1 (very much improved) to 7 (very much worse).
Time Frame: 28 Weeks
Population: The PI has left the institution and this study was terminated due to loss of funding. The data was not analyzed.
Arm/Group | All Participants
Number analyzed (Participants) | 0

5. Secondary Outcome: Computerized Multiphasic Interactive Neurocognitive DualDisplay TM System (CMINDS®)
Time Frame: 28 weeks
Population: The PI has left the institution and this study was terminated due to loss of funding. The data was not analyzed.
Arm/Group | All Participants
Number analyzed (Participants) | 0

6. Secondary Outcome: Mayer-Salovey-Caruso Emotional Intelligence Test: Managing Emotions (MSCEIT™ ME)
Time Frame: 28 Weeks
Population: The PI has left the institution and this study was terminated due to loss of funding. The data was not analyzed.
Arm/Group | All Participants
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | All Participants
All-Cause Mortality (participants affected / at risk) | 0/14
Serious Adverse Events (participants affected / at risk) | 0/14
Other Adverse Events (participants affected / at risk) | 0/14

LIMITATIONS AND CAVEATS:
This study was halted due to an indefinite break in funding. The Principal Investigator has left the institution and there is no way to determine the arms/groups of this study. The study data was never analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes